CLINICAL TRIAL: NCT01760343
Title: A Randomized, Double-blind, Single-center, Cross-over Study to Evaluate the Safety, Bioavailability and Pharmacokinetics of Two Formulations of C1-esterase Inhibitor Administered Intravenously
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of Two Formulations of C1-esterase Inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL830_1001; 2012-002429-31 (EudraCT Number)
Record Dates: First submitted 2012-12-24; First posted 2013-01-04 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Hereditary Angioedema Types I and II
MeSH Terms: conditions — Hereditary Angioedema Types I and II | interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Berinert, then CSL830 (Experimental): A single intravenous dose of Berinert at 1500 units (1500 IU), followed by a single intravenous dose of CSL830 at 1500 IU.
  Interventions: Biological: Berinert; Biological: CSL830
- CSL830, then Berinert (Experimental): A single intravenous dose of CSL830 at 1500 IU, followed by a single intravenous dose of Berinert at 1500 IU.
  Interventions: Biological: Berinert; Biological: CSL830

INTERVENTIONS:
Biological: Berinert — Berinert is a plasma-derived C1 esterase inhibitor (human), supplied as a freeze-dried powder for reconstitution.
Biological: CSL830 — CSL830 is a formulation of Berinert.

SUMMARY:
A new formulation of Berinert (CSL830) is being investigated for the management of hereditary angioedema (HAE). The main aim of the study is to assess the safety of a single 1500 IU dose of the new formulation of Berinert. This study will also look at the pharmacokinetics of CSL830 relative to Berinert currently on the market.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without clinically significant medical conditions or laboratory abnormalities
* Male or female subjects aged 18 to 45 years inclusive, at the time of informed consent
* Non-smokers
* Body mass index of 18.0 to 29.0 kg/m2 inclusive

Exclusion Criteria:

* Previous history of clinically significant arterial or venous thrombosis, current history of a clinically significant pro-thrombotic risk, or a clinically significant abnormality on laboratory thrombotic screen at the screening visit.
* Known or suspected hypersensitivity to the investigational medicinal product (IMP), or to any excipients of the IMP.
* Female subjects who started taking or changed dose of any hormonal contraceptive regimen or hormone replacement therapy (ie, estrogen/progesterone containing products) within 3 months before the screening visit.
* Alcohol, drug, or medication abuse within one year before the study.
* Female subjects of childbearing potential (eg, not post-menopausal) either not using, or not willing to use, a medically reliable method of contraception for the entire duration of the study, or have a vasectomized partner, or not sexually abstinent for the entire duration of the study, or not surgically sterile.
* Participation in another clinical study (or use of another IMP) within 30 days (or 5 times the half-life, whichever is longer) before, or during, the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) within 24 hours of CSL830 infusion | From the start of infusion to 24 hours after the end of infusion

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) within 10 days of the CSL830 infusion | From the start of infusion to 10 days after the infusion
Relative bioavailability of CSL830 versus Berinert - Cmax | 240 hours
  Relative bioavailability in terms of maximum concentration (Cmax) of CSL830 versus Berinert
Relative bioavailability of CSL830 versus Berinert - AUC | 240 hours
  Relative bioavailability in terms of area under the curve from timepoint 0 to infinity (AUC0-∞) of CSL830 versus Berinert

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Program Director, Study Director — CSL Behring
Locations (1):
- Study Site, Berlin, Germany